CLINICAL TRIAL: NCT06442644
Title: Live Music in the Intensive Care Unit
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: Region MidtJylland Denmark (Other); Novo Nordisk A/S (Industry); The Royal Conservatory of Music (Other)
Responsible Party: Principal Investigator, Linette Thorn, Specialized intensive care nurse, Aarhus University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1-10-72-66-24
Record Dates: First submitted 2024-05-03; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Stress; Pain
Keywords: Intensive care unit; Live music; Quantitative; Stress; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adult intensive care patients (Other): Live music interventions
  Interventions: Other: Live music in the intensive care unit

INTERVENTIONS:
Other: Live music in the intensive care unit — To test a patient-tailored live music intervention's effect on stress reduction in adult, critically ill patients admitted to the intensive care unit.

SUMMARY:
The goal of this quasi-experimental pre- post test study is to test a patient-tailored live music intervention's effect on stress and pain reduction in adult, critically ill patients admitted to the intensive care unit.

The main question it aims to answer is:

• Does live music reduce stress and pain in adult intensive care patients?

In the pre-post test design, the patients will be their own control. There will be no randomisation. Researchers will compare measurements of heartrate, respiration rate, heartrate variability, blood pressure and pain before and after the live music intervention to see if live music effects these vital parameters.

Participants will listen to live music in their room in the intensive care unit for 5 to 15 minutes.

DETAILED DESCRIPTION:
1. Introduction The intensive care unit (ICU) has been and is still undergoing paradigmatic changes and technological advancements, meaning that an increased number of patients are conscious during their ICU stay and more survive to remember their ICU admission. Patients are admitted to the ICU because they are in urgent need of life saving treatments. However, an ICU admission can be a traumatic experience for patients and their relatives. The ICU patient room is designed with the purpose of promoting advanced care and treatment performed by the healthcare professionals. However, the room leaves little space for positive sensory inputs for the patients and the relatives; rather the environment is a highly technological, noisy, unfamiliar and often frightening experience for the patients and their relatives - memories of this may follow them for years. In this project, the investigators aim to test patient-tailored live music as an intervention to reduce stress and pain for adult ICU patients.
2. Project aim The aim of this study is to test a patient-tailored live music intervention's effect on stress reduction in adult, critically ill patients admitted to the intensive care unit.
3. Design and analysis method The study is a quasi-experimental pre- post test study, with patients being their own control. The pre-post test measurements will be carried out at predefined time points (5 minutes before and 5 minutes after the intervention). Our primary outcome, the HRV, will be measured continuously 5 minutes before the music intervention, during the whole intervention and 5 minutes after the intervention. There will be no randomisation.

   Relevant static calculations will be performed using Stata. Statistical analysis will be supported by a statistician at CONNECT (A data support centre for clinical and genomic data).
4. Music intervention This study will be performed in collaboration with the Royal Academy of Music, Aarhus, Denmark (RAMA) and ICU departments across Central Denmark Region, Aarhus University Hospital being main investigator.

   The musicians have participated in a training programme after which they are able to carry out one-on-one patient-tailored music sessions for adult patients at the ICU carried out in the patient's room.

   Each music intervention comprises three components: 1) A prior briefing by the nurse on the patients' condition relevant for the musical practice 2) A patient-tailored live music session in the patient room and 3) A debriefing with the nurse.

   The musicians plan a programme for each intervention day, and the patients will therefore not have the opportunity to choose specific pieces of music. The musicians prepare a mix of relaxing, soothing, familiar and unknown music with low-pitched instruments, e.g., guitar and piano, in a slow tempo (60-80 beats per minute), with a predictable musical structure, rhythm, and tonality, as it has been shown that low-pitched and low-intensity music may be calming and may regulate arousal levels. The length of the music intervention will range from 5 to 15 minutes depending on how many music pieces the patient wants to listen to or based on the nurse's assessment of the patient's condition.
5. Sample size Aarhus University Hospital is the main research centre, but the study is a multi-centre study with participation of the Regional Hospitals of Gødstrup, Horsens and Viborg; all have agreed to participate. The intervention is fully implemented at all hospitals.

   The sample size is calculated based on an estimated population of 1103, corresponding to the patients receiving the intervention at all four sites annually. The investigators have determined that a sample size of 202 is needed to estimate the effect with a confidence level of 95%, margin of error of 5% and population proportion of 80%.

   Patients will be included consecutively.
6. Project organisation and feasibility As Aarhus University Hospital is the main study site and also the largest, the investigators will include the majority of patients. This means that the investigators will have a larger percentage of the total sample size than the regional hospitals. A project nurse will collect data at each site.

   The project group consists of one project nurse and one nurse manager at each site.

   Furthermore, the group consists of Professor in Nursing at Aarhus University Hospital Pia Dreyer, Associate Professor at The Royal Academy of Music (Aarhus/Aalborg) Margrethe Langer Bro, project nurse Linette Thorn and the main applicant. The results from this pretest-posttest study will be published in a peer-reviewed journal (e.g., Nursing in Critical Care). Results will also be presented at national and international conferences.
7. Impact of the project Instead of being exposed to an unpleasant room with little opportunity to rest their minds, patients (together with their relatives) will be given the opportunity to experience positive, musical stimuli that bring pleasant experiences and memories, which may support the patients mental well-being and rehabilitation both in the short and long term. The project has the potential to be implemented in more ICU departments across Denmark and potentially also in a broad range of non-ICU hospital departments.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years)
* Admitted to one of the four participating ICU departments for a minimum of 24 hours
* Able to read and speak Danish
* For incapable patients, it is necessary to have a close relative (e.g., spouse or adult child), as these will provide proxy consent for study participation

Exclusion Criteria:

* Unstable patients with a need of change/adjustment of the ongoing treatment of e.g. drug infusions or ventilator settings during the music intervention, as this can possibly affect the HRV measurements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Heartrate variability | baseline (10 minutes before listening to live music), during (5-15 minutes of listening to live music), after (10 minutes after listening to live music)
  measured via the HeartMath Sensor, which is validated for measuring stress levels

SECONDARY OUTCOMES:
Heartrate | baseline (5 minutes before listening to live music), after (5 minutes after listening to live music)
  Heart beat per minut
The patient's subjective pain experience via a numerical ranking scale (NRS) | baseline (5 minutes before listening to live music), after (5 minutes after listening to live music)
  Monitoring pain on a scale of 0-10, where 0 is no pain and 10 is the worst pain imaginable
Patient's self-reported stress level measured by STAI (State-Trait Anxiety Inventory) a validated short version to measure the stress level. | baseline (5 minutes before listening to live music), after (5 minutes after listening to live music)
  Questionaire
Blood pressure | baseline (5 minutes before listening to live music), after (5 minutes after listening to live music)
  Mean arteriel blood pressure meassured by artery cannula
Respiration rate | baseline (5 minutes before listening to live music), after (5 minutes after listening to live music)
  Breaths per minut

CONTACTS AND LOCATIONS:
Overall Officials: Linette Thorn, Master, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Central Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No